CLINICAL TRIAL: NCT04260412
Title: The Effect of Combining Medium Cut Off Polyarylethersulfone-polyvinylpyrrolidone Dialysis Membrane and Diet Modification on Reducing of Inflammation Response
Brief Title: The Effect of Combining Medium Cut Off Dialysis Membrane and Diet Modification on Reducing of Inflammation Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Jernej Pajek, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIIDINFLAMMATION
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: End Stage Renal Disease; Haemodialysis; Diet, Healthy; Chronic Inflammation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Psyllium; sodium propionate

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, interventional, two parallel arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm - MCO dialysis membrane (Experimental): 4 weeks of dialysis with MCO membrane, then dialysis for 4 weeks with MCO membrane and increased fiber intake
  Interventions: Device: medium cut-off (MCO) dialysis membrane; Dietary Supplement: Dietary fiber mixture (Plantago Psyllium 69% and Inulin 30%); Dietary Supplement: Sodium propionate
- Control arm - high-flux membrane haemodiafiltration (Active Comparator): 4 weeks of high-flux membrane haemodiafiltration and 4 weeks of high-flux membrane haemodiafiltration and increased fiber intake
  Interventions: Dietary Supplement: Dietary fiber mixture (Plantago Psyllium 69% and Inulin 30%); Dietary Supplement: Sodium propionate

INTERVENTIONS:
Device: medium cut-off (MCO) dialysis membrane — Medium cut-off dialysis (MCO) membrane is a dialysis membrane with a higher molecular weight retention onset and similar cut-off as standard high-flux dialysis membranes. It is capable of providing increased clearance of medium sized uremic toxins and some plasma proteins (cytokines, inflammatory mediators).
  Other Names: Theranova dialysis membrane (Baxter AG)
  Arms: Interventional arm - MCO dialysis membrane
Dietary Supplement: Dietary fiber mixture (Plantago Psyllium 69% and Inulin 30%) — Dietary fiber (Psyllium 69% and Inulin 30% mixture) added to the meals in the dose of 5g BID for 4 weeks in the second phase of the study.
  Other Names: Kolon3Aktiv (Topnatur s.r.o., Czech republic)
Dietary Supplement: Sodium propionate — Sodium propionate (a short-chain fatty acid) added to the meals in the dose of 500 mg BID in the second phase in the study.

SUMMARY:
The investigators purpose is to research the impact of the simultaneous use of a new dialysis membrane with higher permeability for medium and protein bound uraemic toxins (medium cut-off dialysis membrane Theranova®) combined with diet modification to reduce the level of inflammation in chronic dialysis patients. The investigators hypothesize that the use of a medium-cut off dialysis membrane and dietary modification work synergistically and cause a significant and clinically meaningful reduction in inflammation levels compared to on-line hemodiafiltration with a high-flux dialysis membrane.

DETAILED DESCRIPTION:
The investigators will carry out a prospective interventional randomised study to compare achieved serum concentrations of selected protein bound uremic toxins by dialysis with a medium cut-off membrane (Theranova, Baxter AG, USA) and online hemodiafiltration with a standard "high-flux" dialysis membrane. In the second phase, both dialysis purification methods will be supplemented by a change in the diet with increase of the daily intake of dietary fiber to 30g and addition of a short-chain fatty acid propionate in the dose of 1 g daily.

The main outcome of the study is the serum concentration of Interleukin-6. Secondary outcome is the serum concentration of interleukin-10, serum amyloid A, High-sensitivity C-reactive protein, total leukocyte count and plasma concentration of bacterial 16s rDNA. Serum albumin concentration and lean body weight of patients represent safety outcomes for this study.

This investigator-initiated research project has been entirely planned and will be conducted by the clinical researchers in a tertiary hospital University Medical Center Ljubljana.

The study will include 50 chronic prevalent stable dialysis patients in the following periods:

* 2 weeks of wash-in period with standard bicarbonate haemodialysis and standard high-flux dialysis membrane,
* then the patients will be randomized in a 1:1 ratio to either one of the two study arms:
* (interventional study arm) 4 weeks of dialysis with medium cut-off (Theranova) membrane (first phase), then dialysis for 4 weeks with the same membrane and increased fiber intake (second phase),
* (control study arm) 4 weeks of dialysis with a high-flux membrane using on-line haemodiafiltration (first phase) and 4 weeks of high-flux membrane haemodiafiltration and increased fiber intake (second phase),
* finally, all patients will undergo a 4 week wash-out period with a standard bicarbonate haemodialysis using standard high-flux dialysis membrane identical to wash-in period.

Measurement of the study end-points will be carried out at the end of 2-week wash-in period, each 4-week period and at the end of 4 week wash-out period.

ELIGIBILITY:
Inclusion Criteria:

* Patient on chronic hemodialysis or hemodiafiltration for at least 12 weeks;
* Age 18 years old or more;
* A functioning arteriovenous fistula or graft as a permanent dialysis vascular access;
* Being able to give an informed consent to participate in the survey

Exclusion Criteria:

* Planned kidney transplantation, transition to peritoneal dialysis or to another dialysis center within 12 weeks of the start of the study
* Acute febrile inless 4 weeks prior to study inclusion
* Active chronic inflammation (e.g., an active autoimmune disease or an open wound), chronic ongoing infection or cancer
* New cardiovascular or cerebrovascular event 4 weeks prior to study inclusion
* Clinically malnourishet patient and/or BMI below 19 kg/m2 and/or loss of more the 5% of body mass in the last 3 months
* Immunosuppressive treatment
* Expected survival of less than 1 year
* Pregnancy or breast-feeding
* Indication for dietary supplements to increase calorie and/or protein intake
* Specific indication for carrying out hemodiafiltration instead of hemodialysis as per attending physician
* Serum albumin concentration <32 g/l after screening to enter the study
* Inability to follow the study diet or test procedures
* Rapid reduction of residual renal function in the period prior to entry into the study
* Intolerant of on-line haemodiafiltration (infusion intolerance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Serum concentration of inflammatory mediator interleukin-6 (IL-6). | At the end of wash-in period (basal sample-baseline), at the end of first phase (4 weeks after baseline), at the end of second phase (8 weeks after baseline), at the end of wash-out period (12 weeks after baseline).
  Blood for the laboratory measurements of serum total interleukin-6 concentration will be taken from the arterial line before the start of midweek hemodialysis procedure.

SECONDARY OUTCOMES:
Serum concentration of inflammatory mediator High-sensitivity C-reactive protein (hs-CRP). | At the end of wash-in period (basal sample-baseline), at the end of first phase (4 weeks after baseline), at the end of second phase (8 weeks after baseline), at the end of wash-out period (12 weeks after baseline).
  Blood for the laboratory measurements of serum total hs-CRP concentration will be taken from the arterial line before the start of midweek hemodialysis procedure.

OTHER OUTCOMES:
Serum concentration of inflammatory mediator interleukin-10 (IL-10). | At the end of wash-in period (basal sample-baseline), at the end of first phase (4 weeks after baseline), at the end of second phase (8 weeks after baseline), at the end of wash-out period (12 weeks after baseline).
  Blood for the laboratory measurements of serum total interleukin-10 concentration will be taken from the arterial line before the start of midweek hemodialysis procedure.
Serum concentration of inflammatory mediator serum amyloid A (SAA). | At the end of wash-in period (basal sample-baseline), at the end of first phase (4 weeks after baseline), at the end of second phase (8 weeks after baseline), at the end of wash-out period (12 weeks after baseline).
  Blood for the laboratory measurements of total seum amyloid A concentration will be taken from the arterial line before the start of midweek hemodialysis procedure.
Serum leukocyte count. | At the end of wash-in period (basal sample-baseline), at the end of first phase (4 weeks after baseline), at the end of second phase (8 weeks after baseline), at the end of wash-out period (12 weeks after baseline).
  Blood for the laboratory measurements of total serum leukocyte count will be taken from the arterial line before the start of midweek hemodialysis procedure.
Plasma concentration of bacterial 16s rDNA. | At the end of wash-in period (basal sample-baseline), at the end of first phase (4 weeks after baseline), at the end of second phase (8 weeks after baseline), at the end of wash-out period (12 weeks after baseline).
  Blood for the laboratory measurements of plasma concentration of bacterial 16s rDNA will be taken from the arterial line before the start of midweek hemodialysis procedure.
Serum albumin concentration. | At the end of wash-in period (basal sample-baseline), at the end of first phase (4 weeks after baseline), at the end of second phase (8 weeks after baseline), at the end of wash-out period (12 weeks after baseline).
  Blood for the laboratory measurements of serum albumin concentration will be taken from the arterial line before the start of midweek hemodialysis procedure.
Dialysis symptom index questionnaire score. | At the end of wash-in period (basal sample-baseline), at the end of first phase (4 weeks after baseline), at the end of second phase (8 weeks after baseline), at the end of wash-out period (12 weeks after baseline).
  A validated questionnaire of 30 questions regarding the dialysis symptoms experienced during the last week.
Time to finish 10 repetition sit to stand test. | At the end of wash-in period (basal sample-baseline), at the end of first phase (4 weeks after baseline), at the end of second phase (8 weeks after baseline), at the end of wash-out period (12 weeks after baseline).
  This validated test measures lower limb strength. Participants are required to stand up and sit down 10 times from an armless chair as quickly as possible, the outcome is the time needed to perform the test.
Physical activity level as measured by accelerometry. | At the end of wash-in period (basal sample-baseline), at the end of first phase (4 weeks after baseline), at the end of second phase (8 weeks after baseline), at the end of wash-out period (12 weeks after baseline).
  Number of accelerometer counts in 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jernej Pajek, MD, PhD, Study Chair — Nephrology department, University Medical Centre Ljubljana, Slovenia
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Plan to share IPD that underline results published in the manuscripts reporting study results.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From the time of publication of associated manuscripts for 10 years.
Access Criteria: Available on demand from the investigators.

REFERENCES:
- [Background] Dobre M, Meyer TW, Hostetter TH. Searching for uremic toxins. Clin J Am Soc Nephrol. 2013 Feb;8(2):322-7. doi: 10.2215/CJN.04260412. Epub 2012 Sep 27. PMID 23024165
- [Background] Depner TA. Uremic toxicity: urea and beyond. Semin Dial. 2001 Jul-Aug;14(4):246-51. doi: 10.1046/j.1525-139x.2001.00072.x. PMID 11489197
- [Background] Mostovaya IM, Blankestijn PJ, Bots ML, Covic A, Davenport A, Grooteman MP, Hegbrant J, Locatelli F, Vanholder R, Nube MJ; EUDIAL1 - an official ERA-EDTA Working Group. Clinical evidence on hemodiafiltration: a systematic review and a meta-analysis. Semin Dial. 2014 Mar;27(2):119-27. doi: 10.1111/sdi.12200. PMID 24738146
- [Background] Wang AY, Ninomiya T, Al-Kahwa A, Perkovic V, Gallagher MP, Hawley C, Jardine MJ. Effect of hemodiafiltration or hemofiltration compared with hemodialysis on mortality and cardiovascular disease in chronic kidney failure: a systematic review and meta-analysis of randomized trials. Am J Kidney Dis. 2014 Jun;63(6):968-78. doi: 10.1053/j.ajkd.2014.01.435. Epub 2014 Mar 28. PMID 24685515
- [Background] Zweigart C, Boschetti-de-Fierro A, Hulko M, Nilsson LG, Beck W, Storr M, Krause B. Medium cut-off membranes - closer to the natural kidney removal function. Int J Artif Organs. 2017 Jul 5;40(7):328-334. doi: 10.5301/ijao.5000603. Epub 2017 May 26. No abstract available. PMID 28574113
- [Background] Zickler D, Schindler R, Willy K, Martus P, Pawlak M, Storr M, Hulko M, Boehler T, Glomb MA, Liehr K, Henning C, Templin M, Trojanowicz B, Ulrich C, Werner K, Fiedler R, Girndt M. Medium Cut-Off (MCO) Membranes Reduce Inflammation in Chronic Dialysis Patients-A Randomized Controlled Clinical Trial. PLoS One. 2017 Jan 13;12(1):e0169024. doi: 10.1371/journal.pone.0169024. eCollection 2017. PMID 28085888
- [Background] Eloot S, Van Biesen W, Glorieux G, Neirynck N, Dhondt A, Vanholder R. Does the adequacy parameter Kt/V(urea) reflect uremic toxin concentrations in hemodialysis patients? PLoS One. 2013 Nov 13;8(11):e76838. doi: 10.1371/journal.pone.0076838. eCollection 2013. PMID 24236005
- [Background] Montemurno E, Cosola C, Dalfino G, Daidone G, De Angelis M, Gobbetti M, Gesualdo L. What would you like to eat, Mr CKD Microbiota? A Mediterranean Diet, please! Kidney Blood Press Res. 2014;39(2-3):114-23. doi: 10.1159/000355785. Epub 2014 Jul 29. PMID 25117687
- [Background] Sirich TL. Dietary protein and fiber in end stage renal disease. Semin Dial. 2015 Jan-Feb;28(1):75-80. doi: 10.1111/sdi.12315. Epub 2014 Oct 16. PMID 25319504
- [Background] Claro LM, Moreno-Amaral AN, Gadotti AC, Dolenga CJ, Nakao LS, Azevedo MLV, de Noronha L, Olandoski M, de Moraes TP, Stinghen AEM, Pecoits-Filho R. The Impact of Uremic Toxicity Induced Inflammatory Response on the Cardiovascular Burden in Chronic Kidney Disease. Toxins (Basel). 2018 Sep 23;10(10):384. doi: 10.3390/toxins10100384. PMID 30249039
- [Background] Barrajon-Catalan E, Herranz-Lopez M, Joven J, Segura-Carretero A, Alonso-Villaverde C, Menendez JA, Micol V. Molecular promiscuity of plant polyphenols in the management of age-related diseases: far beyond their antioxidant properties. Adv Exp Med Biol. 2014;824:141-59. doi: 10.1007/978-3-319-07320-0_11. PMID 25038998
- [Background] Moe SM, Zidehsarai MP, Chambers MA, Jackman LA, Radcliffe JS, Trevino LL, Donahue SE, Asplin JR. Vegetarian compared with meat dietary protein source and phosphorus homeostasis in chronic kidney disease. Clin J Am Soc Nephrol. 2011 Feb;6(2):257-64. doi: 10.2215/CJN.05040610. Epub 2010 Dec 23. PMID 21183586
- [Background] Marzocco S, Fazeli G, Di Micco L, Autore G, Adesso S, Dal Piaz F, Heidland A, Di Iorio B. Supplementation of Short-Chain Fatty Acid, Sodium Propionate, in Patients on Maintenance Hemodialysis: Beneficial Effects on Inflammatory Parameters and Gut-Derived Uremic Toxins, A Pilot Study (PLAN Study). J Clin Med. 2018 Sep 30;7(10):315. doi: 10.3390/jcm7100315. PMID 30274359
- [Background] Kirsch AH, Lyko R, Nilsson LG, Beck W, Amdahl M, Lechner P, Schneider A, Wanner C, Rosenkranz AR, Krieter DH. Performance of hemodialysis with novel medium cut-off dialyzers. Nephrol Dial Transplant. 2017 Jan 1;32(1):165-172. doi: 10.1093/ndt/gfw310. PMID 27587605
- [Background] Krishnasamy R, Hawley CM, Jardine MJ, Roberts MA, Cho YJ, Wong MG, Heath A, Nelson CL, Sen S, Mount PF, Pascoe EM, Darssan D, Vergara LA, Paul-Brent PA, Toussaint ND, Johnson DW, Hutchison CA. Design and methods of the REMOVAL-HD study: a tRial Evaluating Mid cut-Off Value membrane clearance of Albumin and Light chains in HaemoDialysis patients. BMC Nephrol. 2018 Apr 17;19(1):89. doi: 10.1186/s12882-018-0883-8. PMID 29665795
- [Background] Borges NA, Barros AF, Nakao LS, Dolenga CJ, Fouque D, Mafra D. Protein-Bound Uremic Toxins from Gut Microbiota and Inflammatory Markers in Chronic Kidney Disease. J Ren Nutr. 2016 Nov;26(6):396-400. doi: 10.1053/j.jrn.2016.07.005. PMID 27751361
- [Background] Chapdelaine I, de Roij van Zuijdewijn CL, Mostovaya IM, Levesque R, Davenport A, Blankestijn PJ, Wanner C, Nube MJ, Grooteman MP; EUDIAL Group; Blankestijn PJ, Davenport A, Basile C, Locatelli F, Maduell F, Mitra S, Ronco C, Shroff R, Tattersall J, Wanner C. Optimization of the convection volume in online post-dilution haemodiafiltration: practical and technical issues. Clin Kidney J. 2015 Apr;8(2):191-8. doi: 10.1093/ckj/sfv003. Epub 2015 Feb 16. PMID 25815176
- [Background] Pajek J, Kveder R, Bren A, Gucek A, Ihan A, Osredkar J, Lindholm B. Short-term effects of a new bicarbonate/lactate-buffered and conventional peritoneal dialysis fluid on peritoneal and systemic inflammation in CAPD patients: a randomized controlled study. Perit Dial Int. 2008 Jan-Feb;28(1):44-52. PMID 18178947